CLINICAL TRIAL: NCT06062316
Title: Early Warning Model of Myocardial Remodeling After Acute Myocardial Infarction Based on Multimodal Feature Structure Technology
Brief Title: Warning Model of Myocardial Remodeling After Acute Myocardial Infarction Using Multimodal Feature Structure Technology
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: xuanwuliuzhi
Record Dates: First submitted 2023-09-17; First posted 2023-10-02 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2023-10

CONDITIONS: Myocardial Infarction
Keywords: Computer aided diagnosis; Myocardial Remodeling; Early warning model; Myocardial infarction; MRI
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute myocardial infarction (AMI) is one of the most important diseases threatening human life. The existing MI prognosis prediction scales mostly predict the incidence of death, recurrent MI and heart failure through 6-8 clinical text indicators, and the data are collected relatively simply. Myocardial remodeling, as an adverse pathological change that can start and continue to progress in the early stage after myocardial infarction, is the main pathological mechanism of heart failure and death. However, there is no quantitative early-warning model of myocardial remodeling, and the clinical guidance of early intervention is lacking.

Our previous study found that cardiac magnetic resonance imaging can accurately quantify the necrotic area and recoverable myocardium in the edematous myocardium after myocardial infarction. In this study, machine learning algorithm, variable convolution network (DCN) and capsule network (capsnet) are used to build a new neural network architecture. Structural feature extraction of multi-modal clinical image data such as MRI and ultrasound is realized. Combined with the established database of 3000 patients with myocardial infarction, the multimodal feature matrix will be constructed, and a variety of classifiers such as support vector machine (SVM) and random forest (RF) will be used for quantitative prediction of myocardial remodeling, and the effects of different classifiers were evaluated. It is expected that this project will establish a quantitative early warning model of myocardial remodeling after acute myocardial infarction in line with the characteristics of Chinese people. The same type of data outside the database will be used for verification to establish an efficient and stable early warning model.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with acute myocardial infarction, aged 18-80 years; 2.The time from onset to treatment is less than 72h 3.Myocardial enzyme Tni/Tnt(+).

Exclusion Criteria:

* 1.Patients with malignant tumors; 2.Patients who could not receive conventional treatment 3.Patients who did not receive coronary angiography, lacking anatomical and imaging data; 4.Patients who have undergone cardiac surgery (except coronary artery bypass surgery)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Criteria for the diagnosis of acute myocardial infarction:
  increased or decreased cardiac biomarkers (preferably cTn), at least once exceeding the 99th percentile of the upper reference value, cut-off variability ≤10%, and at least one evidence of myocardial ischemia (including symptoms, electrocardiographic ischemic changes, pathological Q-waves, or imaging evidence).
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Novel convolutional neural network algorithm and cardiac magnetic resonance imaging to evaluate the occurrence of myocardial remodeling.remodeling after myocardial infarction. | 1year
  (Quantitative characterization of myocardial remodeling, cardiac magnetic resonance imaging quantifying necrotic areas and recoverable myocardium within the edematous myocardium after myocardial infarction).

SECONDARY OUTCOMES:
The multi-dimensional indexes of existing database were compared with the location and course of myocardial remodeling by artificial intelligence method Degree of correlation analysis. | 1year
  Through the new Deformable Convolutional Capsule network that has been developed The Networks (DCCN) study focused on the existing clinical and imaging comprehensive database of patients with acute myocardial infarction Machine learning was performed on the data to complete the extraction of relevant features and logical relationship analysis of myocardial remodeling after myocardial infarction.
  Strong correlation features were screened.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Liu, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Xicheng, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moran AE, Forouzanfar MH, Roth GA, Mensah GA, Ezzati M, Murray CJ, Naghavi M. Temporal trends in ischemic heart disease mortality in 21 world regions, 1980 to 2010: the Global Burden of Disease 2010 study. Circulation. 2014 Apr 8;129(14):1483-92. doi: 10.1161/CIRCULATIONAHA.113.004042. Epub 2014 Feb 26. PMID 24573352
- [Background] Abuomara HZA, Hassan OM, Rashid T, Baraka M. Myocardial performance index as an echocardiographic predictor of early in-hospital heart failure during first acute anterior ST-elevation myocardial infarction. Egypt Heart J. 2018 Jun;70(2):71-75. doi: 10.1016/j.ehj.2017.12.001. Epub 2017 Dec 24. PMID 30166885
- [Background] Hausenloy DJ, Yellon DM. Myocardial ischemia-reperfusion injury: a neglected therapeutic target. J Clin Invest. 2013 Jan;123(1):92-100. doi: 10.1172/JCI62874. Epub 2013 Jan 2. PMID 23281415
- [Background] Hendriks T, Schurer RAJ, Al Ali L, van den Heuvel AFM, van der Harst P. Left ventricular restoration devices post myocardial infarction. Heart Fail Rev. 2018 Nov;23(6):871-883. doi: 10.1007/s10741-018-9711-2. PMID 29770903
- [Background] Iborra-Egea O, Galvez-Monton C, Roura S, Perea-Gil I, Prat-Vidal C, Soler-Botija C, Bayes-Genis A. Mechanisms of action of sacubitril/valsartan on cardiac remodeling: a systems biology approach. NPJ Syst Biol Appl. 2017 Apr 18;3:12. doi: 10.1038/s41540-017-0013-4. eCollection 2017. PMID 28649439
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Seferovic PM, Fragasso G, Petrie M, Mullens W, Ferrari R, Thum T, Bauersachs J, Anker SD, Ray R, Cavusoglu Y, Polovina M, Metra M, Ambrosio G, Prasad K, Seferovic J, Jhund PS, Dattilo G, Celutkiene J, Piepoli M, Moura B, Chioncel O, Ben Gal T, Heymans S, Jaarsma T, Hill L, Lopatin Y, Lyon AR, Ponikowski P, Lainscak M, Jankowska E, Mueller C, Cosentino F, Lund LH, Filippatos GS, Ruschitzka F, Coats AJS, Rosano GMC. Heart Failure Association of the European Society of Cardiology update on sodium-glucose co-transporter 2 inhibitors in heart failure. Eur J Heart Fail. 2020 Nov;22(11):1984-1986. doi: 10.1002/ejhf.2026. Epub 2020 Oct 27. PMID 33068051
- [Background] Pasternak B, Ueda P, Eliasson B, Svensson AM, Franzen S, Gudbjornsdottir S, Hveem K, Jonasson C, Wintzell V, Melbye M, Svanstrom H. Use of sodium glucose cotransporter 2 inhibitors and risk of major cardiovascular events and heart failure: Scandinavian register based cohort study. BMJ. 2019 Aug 29;366:l4772. doi: 10.1136/bmj.l4772. PMID 31467044
- [Background] West R, Jones D. Cardiac rehabilitation and mortality reduction after myocardial infarction: the emperor's new clothes? Evidence against cardiac rehabilitation. Heart. 2013 Jul;99(13):911-3. doi: 10.1136/heartjnl-2013-303705. Epub 2013 May 4. PMID 23644409
- [Background] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Background] Milani RV, Lavie CJ. Impact of cardiac rehabilitation on depression and its associated mortality. Am J Med. 2007 Sep;120(9):799-806. doi: 10.1016/j.amjmed.2007.03.026. PMID 17765050
- [Background] Karuzas A, Rumbinaite E, Verikas D, Ptasinskas T, Muckiene G, Kazakauskaite E, Zabiela V, Jurkevicius R, Vaskelyte JJ, Zaliunas R, Zaliaduonyte-Peksiene D. Accuracy of three-dimensional systolic dyssynchrony and sphericity indexes for identifying early left ventricular remodeling after acute myocardial infarction. Anatol J Cardiol. 2019 Jun;22(1):13-20. doi: 10.14744/AnatolJCardiol.2019.02844. PMID 31264652
- [Background] Kagiyama N, Shrestha S, Cho JS, Khalil M, Singh Y, Challa A, Casaclang-Verzosa G, Sengupta PP. A low-cost texture-based pipeline for predicting myocardial tissue remodeling and fibrosis using cardiac ultrasound. EBioMedicine. 2020 Apr;54:102726. doi: 10.1016/j.ebiom.2020.102726. Epub 2020 Apr 6. PMID 32268274
- [Background] Chirinos JA, Sardana M, Ansari B, Satija V, Kuriakose D, Edelstein I, Oldland G, Miller R, Gaddam S, Lee J, Suri A, Akers SR. Left Atrial Phasic Function by Cardiac Magnetic Resonance Feature Tracking Is a Strong Predictor of Incident Cardiovascular Events. Circ Cardiovasc Imaging. 2018 Dec;11(12):e007512. doi: 10.1161/CIRCIMAGING.117.007512. PMID 30562112
- [Background] Ranka S, Reddy M, Noheria A. Artificial intelligence in cardiovascular medicine. Curr Opin Cardiol. 2021 Jan;36(1):26-35. doi: 10.1097/HCO.0000000000000812. PMID 33060388
- [Background] Ahmad T, Lund LH, Rao P, Ghosh R, Warier P, Vaccaro B, Dahlstrom U, O'Connor CM, Felker GM, Desai NR. Machine Learning Methods Improve Prognostication, Identify Clinically Distinct Phenotypes, and Detect Heterogeneity in Response to Therapy in a Large Cohort of Heart Failure Patients. J Am Heart Assoc. 2018 Apr 12;7(8):e008081. doi: 10.1161/JAHA.117.008081. PMID 29650709
- [Background] Motwani M, Dey D, Berman DS, Germano G, Achenbach S, Al-Mallah MH, Andreini D, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow BJ, Cury RC, Delago A, Gomez M, Gransar H, Hadamitzky M, Hausleiter J, Hindoyan N, Feuchtner G, Kaufmann PA, Kim YJ, Leipsic J, Lin FY, Maffei E, Marques H, Pontone G, Raff G, Rubinshtein R, Shaw LJ, Stehli J, Villines TC, Dunning A, Min JK, Slomka PJ. Machine learning for prediction of all-cause mortality in patients with suspected coronary artery disease: a 5-year multicentre prospective registry analysis. Eur Heart J. 2017 Feb 14;38(7):500-507. doi: 10.1093/eurheartj/ehw188. PMID 27252451
- [Background] Tokodi M, Schwertner WR, Kovacs A, Toser Z, Staub L, Sarkany A, Lakatos BK, Behon A, Boros AM, Perge P, Kutyifa V, Szeplaki G, Geller L, Merkely B, Kosztin A. Machine learning-based mortality prediction of patients undergoing cardiac resynchronization therapy: the SEMMELWEIS-CRT score. Eur Heart J. 2020 May 7;41(18):1747-1756. doi: 10.1093/eurheartj/ehz902. PMID 31923316
- [Background] Sanchez-Cabo F, Rossello X, Fuster V, Benito F, Manzano JP, Silla JC, Fernandez-Alvira JM, Oliva B, Fernandez-Friera L, Lopez-Melgar B, Mendiguren JM, Sanz J, Ordovas JM, Andres V, Fernandez-Ortiz A, Bueno H, Ibanez B, Garcia-Ruiz JM, Lara-Pezzi E. Machine Learning Improves Cardiovascular Risk Definition for Young, Asymptomatic Individuals. J Am Coll Cardiol. 2020 Oct 6;76(14):1674-1685. doi: 10.1016/j.jacc.2020.08.017. PMID 33004133
- [Background] Commandeur F, Slomka PJ, Goeller M, Chen X, Cadet S, Razipour A, McElhinney P, Gransar H, Cantu S, Miller RJH, Rozanski A, Achenbach S, Tamarappoo BK, Berman DS, Dey D. Machine learning to predict the long-term risk of myocardial infarction and cardiac death based on clinical risk, coronary calcium, and epicardial adipose tissue: a prospective study. Cardiovasc Res. 2020 Dec 1;116(14):2216-2225. doi: 10.1093/cvr/cvz321. PMID 31853543
- [Background] Than MP, Pickering JW, Sandoval Y, Shah ASV, Tsanas A, Apple FS, Blankenberg S, Cullen L, Mueller C, Neumann JT, Twerenbold R, Westermann D, Beshiri A, Mills NL; MI3 Collaborative. Machine Learning to Predict the Likelihood of Acute Myocardial Infarction. Circulation. 2019 Sep 10;140(11):899-909. doi: 10.1161/CIRCULATIONAHA.119.041980. Epub 2019 Aug 16. PMID 31416346
- [Background] Tan JH, Hagiwara Y, Pang W, Lim I, Oh SL, Adam M, Tan RS, Chen M, Acharya UR. Application of stacked convolutional and long short-term memory network for accurate identification of CAD ECG signals. Comput Biol Med. 2018 Mar 1;94:19-26. doi: 10.1016/j.compbiomed.2017.12.023. Epub 2018 Jan 2. PMID 29358103
- [Background] D'Ascenzo F, De Filippo O, Gallone G, Mittone G, Deriu MA, Iannaccone M, Ariza-Sole A, Liebetrau C, Manzano-Fernandez S, Quadri G, Kinnaird T, Campo G, Simao Henriques JP, Hughes JM, Dominguez-Rodriguez A, Aldinucci M, Morbiducci U, Patti G, Raposeiras-Roubin S, Abu-Assi E, De Ferrari GM; PRAISE study group. Machine learning-based prediction of adverse events following an acute coronary syndrome (PRAISE): a modelling study of pooled datasets. Lancet. 2021 Jan 16;397(10270):199-207. doi: 10.1016/S0140-6736(20)32519-8. PMID 33453782
- [Background] Fernandez-Ruiz I. Machine learning predicts risk in ACS. Nat Rev Cardiol. 2021 Apr;18(4):230. doi: 10.1038/s41569-021-00521-8. No abstract available. PMID 33531699
- [Derived] Wang S, Zhao Y, Zhao Y, Wang Y, Fan Z, Liu Z. Construction and Clinical Relevance of a Predictive Model of Coronary Microcirculatory Dysfunction in Patients With Acute Myocardial Infarction Following Percutaneous Coronary Intervention. Rev Cardiovasc Med. 2025 Jun 30;26(6):38533. doi: 10.31083/RCM38533. eCollection 2025 Jun. PMID 40630444